CLINICAL TRIAL: NCT01564966
Title: Cardiovascular-Renal Consequences of Reducing Renal Mass After Living Kidney Donation
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Yasar Caliskan, Specialist of Nephrology, MD, Istanbul University
Other Study IDs: 20120209; 4369 (Other: Istanbul University Scientific Research Projects)
Record Dates: First submitted 2012-03-25; First posted 2012-03-28 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2012-03

CONDITIONS: Kidney Failure; Hypertension; Albuminuria; Renal Failure; Inflammation; Endothelial Dysfunction
Keywords: transplantation; inflammation; endothelial dysfunction
MeSH Terms: conditions — Renal Insufficiency; Hypertension; Albuminuria; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Living kidney donors: Those who donate kidneys

SUMMARY:
* A reduce in renal mass may result in remnant single nephron hyperfiltration, with associated proteinuria and an accelerated loss of kidney function.
* Live-donor kidney transplantation is generally considered the best choice for patients who have renal failure and are awaiting transplantation, because these kidneys function better than kidneys from deceased donors, and waiting times for deceased-donor transplants are long
* Although several studies have shown that kidney donation has low short-term morbidity and mortality, the data on long-term outcomes are much less complete.
* This study is designed to prospectively evaluate the effects of unilateral nephrectomy on cardiovascular-renal functions of donors after living kidney donation: the development of hypertension, albuminuria, renal failure, inflammatory and endothelial changes.

DETAILED DESCRIPTION:
Renal dysfunction is associated with accelerated cardiovascular disease even when kidney function is only mildly impaired. Besides, even levels of urinary albumin excretion below the accepted threshold for microalbuminuria are associated with increased cardiovascular risk, and the risk increases as the degree of proteinuria rises.

* Live-donor kidney transplantation is generally considered the best choice for patients who have renal failure and are awaiting transplantation, because these kidneys function better than kidneys from deceased donors, and waiting times for deceased-donor transplants are long. Although several studies have shown that kidney donation has low short-term morbidity and mortality, the data on long-term outcomes are much less complete. The short and long term renal functions of donors after kidney donation were much studied and still remain uncertain, the cardiovascular effects of reduction in renal mass in kidney donors is also not clearly known.
* Endothelial dysfunction (ED) is the first step for subsequent development of atherosclerosis, which can help us to assess the cardiovascular changes after kidney donation. Prospectively examining the endothelial consequences of uninephrectomy in donors may provide useful insight into the existence and pathophysiology of cardiovascular disease in donors and, therefore, into how the cardiovascular disease risk associated with renal impairment might eventually be reduced.

ELIGIBILITY:
Inclusion Criteria:

* living kidney donors
* Ages of 18 and 70
* Creatinine clearance at donation > 80 ml/min/1.73 m2

Exclusion Criteria:

* Low (< 80 ml/min/1.73 m2) creatinine clearance at donation
* Diabetes mellitus
* Hypertension
* Valvular heart disease, any prior coronary intervention
* Congestive heart failure (New York Heart Association class II or greater)
* Cardiac arrhythmia
* A history of cerebral infarction or transient ischemic attack
* Active infection or non-infectious overt inflammation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Living kidney donors in Istanbul Faculty of Medicine
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2008-04; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alaattin Yildiz, Professor of Medicine, MD, Study Director — Istanbul University
Locations (1):
- Division of Nephrology, Istanbul Faculty of Medicine, Istanbul University, Istanbul, Turkey (Türkiye)